CLINICAL TRIAL: NCT06205329
Title: Phase I Study on the Safety, Tolerability, Pharmacokinetics, and Food Effect Evaluation of WPV01 and WPV01 Co-administrated Ritonavir in Healthy Subjects
Brief Title: Study of WPV01 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Westlake Pharmaceuticals (Hangzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WPV01-CP-01
Record Dates: First submitted 2023-03-28; First posted 2024-01-16 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Ritonavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- WPV01 Dose 1-4 (Experimental): WPV01 Dose 1-4 or Placebo
  Interventions: Drug: WPV01 Dose 1-4
- WPV01 Dose 5-8 (Experimental): WPV01 Dose 5-8 co-administrated with ritonavir or Placebo
  Interventions: Drug: WPV01 Dose 5-8 and Ritonavir
- WPV01 Dose 9-12 (Experimental): WPV01 Dose 9-12 or Placebo
  Interventions: Drug: WPV01 Dose 9-12
- WPV01 Dose 13-15 (Experimental): WPV01 Dose 13-15 or Placebo
  Interventions: Drug: WPV01 Dose 13-15 and Ritonavir
- WPV01 Dose 16 (Experimental): WPV01 Dose 16(with high fat meal) or WPV01 Dose 16 (fed)
  Interventions: Drug: WPV01 Dose 16

INTERVENTIONS:
Drug: WPV01 Dose 1-4 — WPV01 Dose 1-4 or Placebo on day 1
  Arms: WPV01 Dose 1-4
Drug: WPV01 Dose 5-8 and Ritonavir — WPV01 Dose 5-8 and Ritonavir or Placebo on day 1
  Arms: WPV01 Dose 5-8
Drug: WPV01 Dose 9-12 — WPV01 Dose 9-12 or Placebo from day 1 to day 6
  Arms: WPV01 Dose 9-12
Drug: WPV01 Dose 13-15 and Ritonavir — WPV01 Dose 13-15 and Ritonavir or Placebo from day 1 to day 6
  Arms: WPV01 Dose 13-15
Drug: WPV01 Dose 16 — Cohort 1:WPV01 Dose 16 or Placebo (with high fat meal) Cohort 2:WPV01 Dose 16 or Placebo (fasted)
  Arms: WPV01 Dose 16

SUMMARY:
A Phase I Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of WPV01 and WPV01 Co-administrated With Ritonavir in Healthy Adult Subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects signed an informed consent form with full understanding of the test content, procedure and possible adverse effects
* Chinese healthy male or female subjects between aged from 18 to 45 years
* Subjects must agree to comply with the contraceptive requirements during the trial and for 3 months after the last dose
* Body weight ≥ 50 kg for men and ≥ 45 kg for women and body mass index in the range of 18.0 ~ 28.0 kg/m2 (including 18.0 and 28.0)
* Subjects must be willing to understand and comply with study procedures and limitations, have the ability to complete the trial as planned, and be able to communicate effectively with the investigator

Exclusion Criteria:

* Participants who have special dietary requirements and cannot abide by the provided food
* Pregnant or lactating women; Women who have pregnancy plan 1 month before trail, during trail or within 3 months after last dose; Women with positive serum pregnancy tests at screening or baseline
* Participants who have evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic disease
* Participants who have history of any other acute or chronic illness
* Participants who have known allergy to any ingredient in the study treatment drug
* Participants who are judged by the investigator to be unsuitable to participate in this study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-03-11 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single and multiple oral doses of WPV01 and WPV01 in combination with ritonavir in healthy subjects. | Day 1 to Day 18
  Adverse events, including type, incidence, grade (determined with reference to NCI-CTCAE V5.0)

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) in Single Ascending Dose (SAD) | SAD part: Day 1 to Day 18
  The maximum observed plasma concentration (Cmax) is estimated based on the plasma concentrations
Time for Cmax (Tmax) in SAD | SAD part: Day 1 to Day 18
  Tmax was summarized by dosing regimen. It was observed directly from data as time of first occurrence.
Area Under the Concentration-Time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) in SAD | SAD part: Day 1 to Day 18
  AUClast is summarized by dosing regimen and determined by linear/log trapezoidal method.
Area Under the Plasma Concentration-Time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) in SAD | SAD part: Day 1 to Day 18
  AUCinf = Area under the plasma concentration versus time curve (AUC) from time 0 (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf).
Terminal Elimination Half-Life (t½) in SAD | SAD part: Day 1 to Day 18
  t1/2 is summarized by dosing regimen . It is determined by loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log linear concentration time curve. Only those data points judged to describe the terminal log linear decline is used in the regression.
Apparent Clearance (CL/F) in SAD | SAD part: Day 1 to Day 18
  CL/F is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Calculated as Dose/AUCinf. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) in SAD | SAD part: Day 1 to Day 18
  Vz/F is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vz/F is influenced by the fraction absorbed.
Cmax in Multiple Ascending Dose (MAD) | MAD part: Day 1 to Day 22
  Observed Cmax is estimated based on the plasma concentrations
Time for Cmax (Tmax) in MAD | MAD part: Day 1 to Day 22
  Tmax was summarized by dosing regimen. It was observed directly from data as time of first occurrence.
Area Under the Plasma Concentration-Time Profile From Time Zero To End of Dosing Interval (AUCtau) in MAD | MAD part: Day 1 to Day 22
  AUCtau is summarized by dosing regimen and period. Dosing interval is the interval tau between administration of doses of drug. In this study, the dosing interval is 8 hours for three times daily (TID) dosing and 12 hours for twice daily (BID) dosing. It is determined by linear/log trapezoidal method.
To evaluate the metabolites of single oral doses of WPV01 and WPV01 in combination with ritonavir in healthy subjects | MAD part: Day 1 to Day 22
  Urine and stool samples will be collected for metabolite analysis. The major metabolites will be identified and, if necessary, quantitatively identified.
Cmax in Food Effect (FE) | Day 1 to Day 22
  The maximum observed plasma concentration (Cmax) is estimated based on the plasma concentrations of cohort 1 and cohort 2 in FE part.
Tmax in FE | Day 1 to Day 22
  It was observed directly from data as time of first occurrence in cohort 1 and cohort 2 of FE part.
Area Under the Concentration-Time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) in FE | Day 1to Day 22
  AUClast was summarized using the data in cohort 1 and cohort 2 of FE part.

CONTACTS AND LOCATIONS:
Locations (1):
- Shulan(Hangzhou) Hospital, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided
6 months after summary data has been published, sponsor will share the IPD and additional supporting information after internal approval process.